CLINICAL TRIAL: NCT04619225
Title: Correlation Between Cardiac Output and Recovery Time After Reversal of Rocuronium-Induced Blockade With Sugammadex
Brief Title: Cardiac Output and Recovery Time
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of interest
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, J. Ross Renew, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-001771
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Residual Neuromuscular Blockade
Keywords: Neuromuscular Blockade; Tetragraph; AMG; EMG
MeSH Terms: conditions — Delayed Emergence from Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- TetraGraph monitoring (Experimental): Subject scheduled to undergo an elective surgical procedure will have TetraGraph device lead placement on either hand at a discretion of the anesthesiologist
  Interventions: Device: TetraGraph

INTERVENTIONS:
Device: TetraGraph — FDA approved neuromuscular transmission monitor capable of measuring the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to electrical neurostimulation via skin electrodes.

SUMMARY:
The purpose of this research is to determine the time it takes to reverse the effects of the intraoperative medication given to relax the muscles and how this period of recovery correlates with a function of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Age > or = 18 years old.
* Patients willing to participate and provide an informed consent.
* Patients undergoing an elective surgical procedure requiring administration of rocuronium, and the use of a pulmonary artery catheter intraoperatively.

Exclusion Criteria:

* Patients with unilateral disorders, such as stroke, carpal tunnel syndrome, broken wrist with nerve damage, Dupuytren contracture.
* Patients with systemic neuromuscular diseases such as myasthenia gravis.
* Patients with significant organ dysfunction that can significantly affect pharmacokinetics of neuromuscular blocking and reversal agents, i.e., severe renal impairment or end-stage liver disease.
* Patients having surgery that would involve prepping the arm or leg into the sterile field.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J.Ross Renew, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- TetraGraph Monitoring: Subjects scheduled to undergo an elective surgical procedure had TetraGraph device lead placement on either hand at a discretion of the anesthesiologist
  TetraGraph: FDA approved neuromuscular transmission monitor capable of measuring the depth of neuromuscular block in anesthetized patients who received neuromuscular blocking agents. TetraGraph uses EMG to measure the muscle action potentials that are generated in response to electrical neurostimulation via skin electrodes.
Period: Overall Study
Arm/Group | TetraGraph Monitoring
Started | 7
Completed | 5
Not Completed | 2
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Arm/Group | TetraGraph Monitoring
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 7
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.5 (9.39)

OUTCOME MEASURES:

1. Primary Outcome: Recovery Time After Administration of Sugammadex and Its Correlation to Cardiac Output Measure
Description: The correlation between the mean change in cardiac output measurement after reversal with sugammadex to the time it takes to recover from the rocuronium-induced blockade. The Pearson's correlation method was used to calculate the correlation coefficient.
Time Frame: Up to 1 hour postoperative
Measure: Number (95% Confidence Interval); unit: Correlation Coefficient
Arm/Group | TetraGraph Monitoring
Number analyzed (Participants) | 5
Correlation Coefficient | -0.69 [-0.98 to 0.49]
Statistical Analysis 1: Comparison: TetraGraph Monitoring; Test type: Superiority; p = 0.199, Pearson Correlation Coefficients

2. Secondary Outcome: Correlation of Speed of Recovery From Neuromuscular Blockade and Age.
Description: The correlation between the mean change in the speed of recovery from neuromuscular blockade to participant's age. The Pearson's correlation method was used to calculate the correlation coefficient.
Time Frame: Up to 1 hour postoperative
Measure: Number (95% Confidence Interval); unit: Correlation Coefficient
Arm/Group | TetraGraph Monitoring
Number analyzed (Participants) | 5
Correlation Coefficient | -0.464 [-0.955 to 0.708]
Statistical Analysis 1: Comparison: TetraGraph Monitoring; Test type: Superiority; p = 0.431, Pearson's Correlation Coefficients

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of informed consent through up to 10 minutes after arrival to Post-Anesthesia Care Unit (PACU) or when Train of Four (TOF) ratio was > 0.9 (whichever occurred first).
Description: Adverse events were collected through specific questioning and, as appropriate, by examination.
Arm/Group | TetraGraph Monitoring
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
The study was terminated early due to a lack of interest.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT04619225/Prot_SAP_000.pdf